CLINICAL TRIAL: NCT05321082
Title: A Double Blind, Randomized, Placebo-controlled Trial Evaluating the Efficacy and Safety of BI 1015550 Over at Least 52 Weeks in Patients With Progressive Fibrosing Interstitial Lung Diseases (PF-ILDs)
Brief Title: A Study to Find Out Whether BI 1015550 Improves Lung Function in People With Progressive Fibrosing Interstitial Lung Diseases (PF-ILDs)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1305-0023; 2022-001134-11 (EudraCT Number)
Record Dates: First submitted 2022-04-04; First posted 2022-04-11 (Actual); Results first posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Lung Diseases, Interstitial
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — BI 1015550

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Nerandomilast 9 mg (Experimental): Patients with progressive fibrosing interstitial lung disease (PF-ILD) or progressive pulmonary fibrosis (PPF), other than idiopathic pulmonary fibrosis (IPF), were administered 9 milligrams (mg) nerandomilast, taken orally as film-coated tablets twice daily (18 mg total), in the morning and in the evening for an initial 52 weeks, followed by a variable duration till end of trial.
  Interventions: Drug: BI 1015550
- Nerandomilast 18 mg (Experimental): Patients with progressive fibrosing interstitial lung disease (PF-ILD) or progressive pulmonary fibrosis (PPF), other than idiopathic pulmonary fibrosis (IPF), were administered 18 mg nerandomilast, taken orally as film-coated tablets twice daily (36 mg total), in the morning and in the evening for an initial 52 weeks, followed by a variable duration till end of trial.
  Interventions: Drug: BI 1015550
- Placebo (Placebo Comparator): Patients with progressive fibrosing interstitial lung disease (PF-ILD) or progressive pulmonary fibrosis (PPF), other than idiopathic pulmonary fibrosis (IPF), were administered placebo matching nerandomilast, taken orally as film-coated tablets twice daily, in the morning and in the evening for an initial 52 weeks, followed by a variable duration till end of trial.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 1015550 — Participants received film-coated nerandomilast tablets orally, twice daily, at doses of either 9 mg or 18 mg, in the morning and in the evening.
  Other Names: Nerandomilast, JASCAYD®
  Arms: Nerandomilast 18 mg; Nerandomilast 9 mg
Drug: Placebo — Participants received placebo matching 9 mg or 18 mg nerandomilast film-coated tablets orally, twice daily, in the morning and in the evening.
  Arms: Placebo

SUMMARY:
This study is open to adults with Progressive Fibrosing Interstitial Lung Diseases (PF-ILDs). People who have a form of PF-ILD other than Idiopathic Pulmonary Fibrosis (IPF) can join the study. If they already take nintedanib, they can continue treatment throughout the study.

The purpose of this study is to find out whether a medicine called BI 1015550 helps people with PF-ILD. Participants are put into 3 groups randomly, which means by chance. Participants in 2 groups take different doses of BI 1015550 as tablets twice a day. Participants in the placebo group take placebo tablets twice a day. Placebo tablets look like BI 1015550 tablets but do not contain any medicine.

Participants are in the study for up to two and a half years. During the first year, they visit the study site 10 times. Afterwards, they visit the study site every 3 months. The doctors regularly test participants' lung function. The results of the lung function tests are compared between the groups. The doctors also regularly check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion criteria

1. Patients ≥18 years old at the time of signed informed consent.
2. Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial.
3. Diagnosis of progressive fibrosing ILD other than IPF (physician confirmed).
4. Patients may be either:

   * on a stable therapy* with nintedanib for at least 12 weeks prior to Visit 1 and during screening and are planning to stay on this background treatment after randomization. (*stable therapy is defined as a tolerated regimen of nintedanib (with no dose changes) for at least 12 weeks)
   * not on treatment with nintedanib for at least 8 weeks prior to Visit 1 and during the screening period (e.g. either Antifibrotic (AF)-treatment naïve or previously discontinued) and do not plan to start or re-start antifibrotic treatment.
5. Forced Vital Capacity (FVC) ≥45% of predicted normal at Visit 1.
6. DLCO ≥25% of predicted normal corrected for hemoglobin (Hb) at Visit 1.
7. Women of childbearing potential (WOCBP) must be ready and able to use highly effective methods of birth control. WOCBP taking oral contraceptives (OCs) also have to use one barrier method
8. Patients treated with permitted immunosuppressive agents (other than corticosteroids) for an underlying systemic disease (e.g. Methotrexate (MTX), Azathioprine (AZA)) need to be on a stable treatment for at least 12 weeks prior to Visit 1 and during the screening period.

Exclusion criteria

1. Prebronchodilator Forced Expiratory Volume in 1 second (FEV1)/Forced vital capacity (FVC) <0.7 at Visit 1
2. In the opinion of the Investigator, other clinically significant pulmonary abnormalities.
3. Acute Interstitial Lung Disease (ILD) exacerbation within 3 months prior to Visit 1 and/or during the screening period (investigator-determined).
4. Relevant chronic or acute infections including human immunodeficiency virus (HIV) and viral hepatitis.
5. Patients having developed ILD due to severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection/coronavirus disease 2019 (COVID-19) within 12 months of screening (based on investigators judgement).
6. Major surgery (major according to the investigator's assessment) performed within 6 weeks prior to Visit 2 or planned during the trial period, e.g. hip replacement. Registration on lung transplantation list would not be considered as planned major surgery.
7. Any documented active or suspected malignancy or history of malignancy within 5 years prior to Visit 1, except appropriately treated basal cell carcinoma of the skin, in situ squamous cell carcinoma of the skin or in situ carcinoma of uterine cervix.
8. Aspartate aminotransferase (AST) or Alanine Aminotransferase (ALT) >2.5 x upper limit of normal (ULN) or total Bilirubin >1.5 x ULN at Visit 1.

Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1178 (Actual)
Dates: Start 2022-11-16 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2025-04-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (400):
- United States (59):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Arizona, Tucson, Arizona
  - University of Southern California, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - University of California Davis, Sacramento, California
  - National Jewish Health, Denver, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Christiana Hospital, Newark, Delaware
  - St. Francis Medical Institute, Clearwater, Florida
  - University of Florida Health Shands Hospital, Gainesville, Florida
  - Clinical Research Specialists LLC, Kissimmee, Florida
  - Advanced Pulmonary Research Institute, Loxahatchee Groves, Florida
  - Destin Pulmonary Critical Care, Santa Rosa Beach, Florida
  - Piedmont Physicians Pulmonary & Sleep Medicine of Buckhead, Atlanta, Georgia
  - The Emory Clinic, Atlanta, Georgia
  - Evanston Hospital Pulmonary Clinic, Evanston, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Tulane University Hospital and Clinic, New Orleans, Louisiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - St. Elizabeth's Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Infinity Medical Research, North Dartmouth, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Beaumont Health, Royal Oak, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Renown Regional Medical Center, Reno, Nevada
  - Stony Brook University Medical Center, Commack, New York
  - Lenox Hill Hospital, New York, New York
  - Columbia University Medical Center-New York Presbyterian Hospital, New York, New York
  - NewYork-Presbyterian/Weill Cornell Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Southeastern Research Center-Winston-Salem-61365, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - The Oregon Clinic, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Jefferson Health Honickman Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Infinity Medical Research, Inc., East Providence, Rhode Island
  - Lowcountry Lung and Critical Care, Charleston, South Carolina
  - Clinical Trials Center of Middle Tennessee, LLC, Franklin, Tennessee
  - Vanderbilt University Medical Center - Vanderbilt Lung Institute at 100 Oaks, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - Premier Pulmonary Critical Care and Sleep Medicine, Denison, Texas
  - UT Health San Antonio, San Antonio, Texas
  - Intermountain Medical Center-Murray-69497, Murray, Utah
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - University of Vermont, Burlington, Vermont
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
- Argentina (10):
  - Centro de Investigaciones Metabolicas (CINME)-C.A.B.A-61553, C.a.b.a
  - CEDIC - Centro de Investigacion Clinica, CABA
  - Hospital Italiano de Buenos Aires, CABA
  - Consultorios Médicos del Buen Ayre, Capital Federal
  - APRILLUS-Asistencia e Investigacion, Ciudad Autonoma Buenos Aires
  - CEMER-Centro Medico De Enfermedades Respiratorias, Florida
  - Instituto Ave Pulmo, Mar del Plata
  - INSARES, Mendoza
  - Centro Respiratorio de Quilmes, Quilmes
  - Instituto Médico de la Fundación Estudios Clínicos, Rosario
- Australia (13):
  - Canberra Hospital, Garran, Australian Capital Territory
  - Royal Prince Alfred Hospital, Camperdown, Sydney, New South Wales
  - Macquarie University, Macquarie Park, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Lung Research Queensland, Chermside, Queensland
  - The Prince Charles Hospital, Chermside, Queensland
  - Mater Hospital Brisbane, South Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Lung Research Victoria, Footscray, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - Trialswest, Spearwood, Western Australia
- Austria (9):
  - Medical University of Graz State Hospital - University Hospital Graz, Graz
  - LKH Klagenfurt am Woerthersee, Klagenfurt
  - Krems University Hospital, Krems
  - Hospital Elisabethinen Linz, Linz
  - LKH Salzburg University Hospital, Salzburg
  - AKH - Medical University of Vienna, Vienna
  - Standort Penzing der Klinik Ottakring, Vienna
  - Clinic Floridsdorf, Vienna
  - Klinikum Wels - Grieskirchen GmbH, Wels
- Belgium (7):
  - Ziekenhuis Netwerk Antwerpen (ZNA) - Campus Middelheim, Antwerp
  - ULB Hopital Erasme, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - UZ Leuven, Leuven
  - Centre Hospitalier Universitaire de Liège, Liège
  - Yvoir - UNIV UCL de Mont-Godinne, Yvoir
- Brazil (11):
  - Serviços Medicos Respirar Sul Fluminense, Barra Mansa
  - Hospital das Clinicas da Universidade Federal de Minas Gerais (HCUFMG), Belo Horizonte,Minas Gerais
  - Edumed - Educacao e Saude SA, Curitiba
  - CLARE - Clinica de Pneumologia, Goiânia
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre, Porto Alegre
  - Hospital Nossa Senhora da Conceição, Porto Alegre - RS
  - Instituto D´Or de Pesquisa e Ensino - Bahia, Salvador
  - Faculdade de Medicina do ABC, Santo André
  - CEMEC - Centro Multidisciplinar de Estudos Clínicos, São Bernardo do Campo
  - Hospital Alemao Oswaldo Cruz, São Paulo
  - Hospital das Clinicas da FMUSP, São Paulo
- Canada (11):
  - Kelowna Respirology & Allergy Research, Kelowna, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - St. Paul's Hospital (Vancouver), Vancouver, British Columbia
  - Dr. Georges-L.-Dumont University Hospital Centre, Moncton, New Brunswick
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Dr. Syed Anees Medicine Professional Corporation, Windsor, Ontario
  - Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec
  - McGill University Health Centre (MUHC), Montreal, Quebec
  - IUCPQ (Laval University), Québec, Quebec
  - CIC Mauricie Inc., Trois-Rivières, Quebec
  - Royal University Hospital (Saskatoon), Saskatoon, Saskatchewan
- Chile (2):
  - Instituto Nacional del Tórax, Providencia, Santiago de Chile
  - Centro de Investigación del Maule, Talca
- China (41):
  - Beijing Chao-Yang Hospital, Beijing
  - China-Japan Friendship Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Chinese PLA General Hospital, Beijing
  - The Second Xiangya Hospital Of Central South University, Changsha
  - West China Hospital of Sichuan University, Chengdu
  - Guangdong Provincial People's Hospital, Guangzhou
  - First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - NanFang Hosptial, Guangzhou
  - Hangzhou First People's Hospital, Hangzhou
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou
  - Zhejiang Hospital, Hangzhou
  - Sir Run Run Shaw Hospital, Zhejiang University, School of Medicine, Hangzhou
  - Anhui Provincial Hospital, Hefei
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot
  - The First hospital of Jiaxing, Jiaxing
  - Jinhua Municipal Central Hospital, Jinhua
  - Nanjing Drum Tower Hospital, Nanjing
  - Ningbo Medical Center Lihuili Hospital, Ningbo
  - The First Affiliated Hospital of Ningbo University, Ningbo
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai
  - Shanghai Chest Hospital, Shanghai
  - Zhongshan Hospital Affiliated to Fudan University, Shanghai
  - Huadong Hospital affiliated to Fudan University, Shanghai
  - Shanghai Pulmonary Hospital, Shanghai
  - China Shenyang Chest Hospital, Shenyang
  - Shenzhen People's Hospital, Shenzhen
  - The University of Hong Kong-Shenzhen Hospital, Shenzhen
  - People's Hospital of Sichuan Province, Sichuan
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Tianjin Medical University General Hospital, Tianjin
  - The First Affiliated Hospital of Wenzhou Medical University, Wenxzhou
  - Wuhan Union Hospital, Wuhan
  - Tongji Hospital Affiliated Tongji Medical College Huazhong University of S & T, Wuhan
  - Renmin Hospital of Wuhan University, Wuhan
  - Wuxi People's Hospital, Wuxi
  - Second Affiliated Hospital of Xi'an JiaoTong University, Xi'an
  - Affiliated Hospital, Xuzhou Medical college, Xuzhou
  - Yichang Central People's Hospital, Yichang
  - General Hospital of Ningxia Medical University, Yinchuan
  - Yuncheng Central Hospital, Yuncheng
- Croatia (3):
  - University hospital center Zagreb, Zagreb
  - University Hospital Dubrava, Zagreb
  - Solmed Polyclinic, Zagreb
- University Thomayer´s Hospital, Prague, Czechia
- Denmark (2):
  - Herlev and Gentofte Hospital, Hellerup
  - Odense University Hospital, Odense
- North Estonia Medical Centre Foundation, Tallinn, Tallinn, Estonia
- Finland (4):
  - HYKS Keuhkosairauksien tutkimusyksikkö, Helsinki
  - Oulun yliopistollinen keskussairaala, Oulu
  - Tampere University Hospital, Tampere
  - TYKS, Turku
- France (22):
  - HOP d'Angers, Angers
  - HOP Avicenne, Bobigny
  - HOP de la Cavale Blanche, Brest
  - HOP Louis Pradel, Bron
  - HOP CHU Caen, Caen
  - HOP François Mitterrand, Dijon
  - HOP Michallon, La Tronche
  - INS Coeur Poumon, Lille
  - HOP Nord, Marseille
  - HOP Arnaud de Villeneuve, Montpellier
  - HOP Nord Laennec, Nantes
  - HOP Pasteur, Nice
  - HOP Européen G. Pompidou, Paris
  - HOP Bichat, Paris
  - HOP Haut-Lévêque, Pessac
  - HOP Robert Debré, Reims
  - HOP Pontchaillou, Rennes
  - HOP Charles Nicolle, Rouen
  - HOP Civil, Strasbourg
  - HOP Foch, Suresnes
  - HOP Larrey, Toulouse
  - HOP Bretonneau, Tours
- Georgia (2):
  - National Center for Tuberculosis and Lung Diseases, Tbilisi, Tbilisi
  - LLC Diacor, Tbilisi
- Germany (21):
  - Velocity Clinical Research Germany GmbH, Ahrensburg, Ahrensburg
  - CIMS Studienzentrum Bamberg GmbH, Bamberg
  - Vivantes Netzwerk für Gesundheit GmbH, Berlin
  - Universitätsklinikum Bonn AöR, Bonn
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Fachkrankenhaus Coswig GmbH, Coswig
  - Ruhrlandklinik, Westdeutsches Lungenzentrum am Universitätsklinikum Essen gGmbH, Essen
  - Universitätsklinikum Hamburg, Eppendorf, Hamburg
  - Klinikum Region Hannover GmbH, Hanover
  - Medizinische Hochschule Hannover, Hanover
  - Thoraxklinik-Heidelberg gGmbH am Universitätsklinikum Heidelberg, Heidelberg
  - Lungenklinik Hemer, Hemer
  - Lungenfachklinik Immenhausen, Immenhausen
  - Klinikum Konstanz, Konstanz
  - Klinikum der Universität München AÖR, München
  - Westfälische Wilhelms-Universität Münster, Münster
  - Klinikum Nürnberg, Nuremberg
  - Krankenhaus Bethanien gGmbH, Solingen
  - Helios Hanseklinikum Stralsund, Stralsund
  - Robert Bosch Gesellschaft für medizinische Forschung mbH, Stuttgart
  - Universitätsklinikum Tübingen, Tübingen
- Greece (5):
  - General Hospital of Athens "Laiko", Athens
  - Hospital of Heraklion (PAGNI), Crete
  - Univ. Gen. Hosp. of Ioannina, Ioannina
  - Univ. Gen. Hosp. of Patras, Pátrai
  - General Hospital of Thessaloniki "Hippokrateio", Thessaloniki
- Hungary (3):
  - Semmelweis University, Budapest
  - Koranyi National Institute For Pulmonolgy, Budapest
  - University of Debrecen Clinical Centre, Debrecen
- India (4):
  - Hindustan Hospital, Coimbatore
  - Bhatia Hospital, Mumbai
  - P.D. Hinduja National Hospital, Mumbai
  - Jehangir Clinical Development Centre Pvt. Ltd., Pune
- Mater Misericordiae University Hospital, Dublin, Ireland
- Israel (5):
  - Shamir Medical Center (Assaf Harofeh), Beer Yaakov
  - Soroka Univ. Medical Center, Beersheba
  - Lady Davis Carmel Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem 91031, Jerusalem
  - Sourasky Medical Center, Tel Aviv
- Italy (16):
  - ASST degli Spedali Civili di Brescia, Brescia
  - A.O.U. Policlinico Vittorio Emanuele, Catania
  - A. O. Universitaria Careggi, Florence
  - Ospedale Colonnello D Avanzo, Foggia
  - Ospedale G.B. Morgagni, Forlì
  - Ospedale San Paolo-MILANO-18793, Milan
  - Ospedale Classificato San Giuseppe, Milan
  - Azienda Ospedaliero-Universitaria di Modena, Modena
  - A.O. San Gerardo di Monza, Monza
  - Osp. dei Colli Monaldi, Napoli
  - Azienda Ospedaliera Universitaria di Padova, Padua
  - Pol. Universitario Tor Vergata, Roma
  - Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma
  - A.O.U. Senese, Siena
  - Ospedali Riuniti di Ancona, Torrette Di Ancona (Ancona)
  - Ospedale di Cattinara, Trieste
- Japan (39):
  - Tosei General Hospital, Aichi, Seto
  - Fujita Health University Hospital, Aichi, Toyoake
  - University of Fukui Hospital, Fukui, Yoshida-gun
  - National Hospital Organization Kyushu Medical Center, Fukuoka, Fukuoka
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Aso Co.,Ltd Iizuka Hospital, Fukuoka, Iizuka
  - Hospital of the University of Occupational and Environmental Health, Fukuoka, Kitakyushu
  - Kurume University Hospital, Fukuoka, Kurume
  - Fukushima Medical University Hospital, Fukushima, Fukushima
  - Tsuboi Hospital, Fukushima, Koriyama
  - Hiroshima Prefectural Hospital, Hiroshima, Hiroshima
  - Sapporo Medical University Hospital, Hokkaido, Sapporo
  - Hokkaido University Hospital, Hokkaido, Sapporo
  - National Hospital Organization Himeji Medical Center, Hyogo, Himeji
  - Kobe City Medical Center General Hospital, Hyogo, Kobe
  - Kobe City Hospital Organization Kobe City Medical Center West Hospital, Hyogo, Kobe
  - Kagawa University Hospital, Kagawa, Kita-gun
  - Kanagawa Cardiovascular and Respiratory Center, Kanagawa, Yokohama
  - Saiseikai Kumamoto Hospital, Kumamoto, Kumamoto
  - Kyoto University Hospital, Kyoto, Kyoto
  - Tohoku University Hospital, Miyagi, Sendai
  - Nagasaki University Hospital, Nagasaki, Nagasaki
  - Kindai University Hospital, Osaka, Sakai
  - National Hospital Organization Kinki-Chuo Chest Medical Center, Osaka, Sakai
  - Osaka Medical and Pharmaceutical University Hospital, Osaka, Takatsuki
  - Saitama Red Cross Hospital, Saitama, Saitama
  - Hamamatsu University Hospital, Shizuoka, Hamamatsu
  - Jichi Medical University Hospital, Tochigi, Shimotsuke
  - Tokushima University Hospital, Tokushima, Tokushima
  - Juntendo University Hospital, Tokyo, Bunkyo-ku
  - Institute of Science Tokyo Hospital, Tokyo, Bunkyo-ku
  - Nippon Medical School Hospital, Tokyo, Bunkyo-ku
  - Toranomon Hospital, Tokyo, Minato-ku
  - Kyorin University Hospital, Tokyo, Mitaka
  - Toho University Omori Medical Center, Tokyo, Ota-ku
  - Tokyo Medical University Hospital, Tokyo, Shinjuku-ku
  - Keio University Hospital, Tokyo, Shinjuku-ku
  - National Center for Global Health and Medicine, Tokyo, Shinjuku-ku
  - Wakayama Medical University Hospital, Wakayama, Wakayama
- Malaysia (4):
  - Hospital Sultan Idris Shah Serdang, Kajang
  - Institut Perubatan Respiratori, Kuala Lumpur
  - Sarawak General Hospital, Kuching
  - Hospital Pulau Pinang-Pulau Pinang-21953, Pulau Pinang
- Mexico (7):
  - Centro de Investigacion Integral MEDIVEST S.C, Chihuahua City
  - CREPID Aire y Salud, Coyoacán
  - Centro de Investigacion Farmacologica del Bajío, S.C., León
  - Soltmed Smo, Mexico City
  - Centro Respiratorio de Mexico, Mexico City
  - Centro de Prevención y Rehabilitación de Enfermedades Pulmon, Monterrey
  - Oaxaca Site Management Organization, S.C., Oaxaca City
- Netherlands (4):
  - Zuyderland Medisch Centrum, Heerlen
  - Leids Universitair Medisch Centrum (LUMC), Leiden
  - St. Antonius ziekenhuis, locatie Nieuwegein, Nieuwegein
  - Erasmus Medisch Centrum-ROTTERDAM-50697, Rotterdam
- New Zealand (4):
  - Waikato Hospital, Hamilton
  - Greenlane Clinical Centre, One Tree Hill, Auckland
  - Middlemore Clinical Trials, Papatoetoe
  - Tauranga Hospital, Tauranga South
- Norway (3):
  - Haukeland Universitetssykehus, Bergen
  - Akershus Universitetssykehus HF, Lørenskog
  - Oslo Universitetssykehus HF, Rikshospitalet, Oslo
- Poland (5):
  - University Clinical Center, Gdansk, Gdansk
  - Leszek Giec Upper-Silesian Med.Cent.Silesian Med.Univ., Katowice
  - Alergopneuma Medical Center, Świdnik
  - Nat.Instit.of Tuberculosis&LungDiseases,Outpat.Clin,warszawa, Warsaw
  - University Clinical Center of the Medical University of Warsaw, Warsaw
- Portugal (4):
  - ULS Braga, Braga
  - ULS de São José, E.P.E., Lisbon
  - USLM, EPE - Hospital Pedro Hispano, Matosinhos Municipality
  - ULS de Gaia/Espinho, EPE, Vila Nova de Gaia
- Allianze Pulmonary Research LLC, Guaynabo, Puerto Rico
- Saudi Arabia (3):
  - King Fahad Specialist Hospital - Research Center, Dammam
  - King Faisal Specialist Hospital and Research Center, Riyadh
  - King Abdullah International Medical Research Center, Riyadh
- Serbia (4):
  - University Clinical Center of Serbia, Belgrade
  - Institute for Pulmonary Diseases of Vojvodina, Kamenitz
  - University Clinical Center of Kragujevac, Kragujevac
  - University Clinical Center Nis, Niš
- Singapore (2):
  - National University Hospital-Singapore-42005, Singapore
  - Singapore General Hospital, Singapore
- Hospital Golnik - Univ. Clinic of Pulmonary and Allergic Diseases, Golnik, Slovenia
- South Africa (3):
  - Busamed Paardevlei Private Hospital, Cape Town
  - Melomed Gatesville Hospital, Cape Town
  - KwaPhila Health Solutions, Durban
- South Korea (8):
  - The Catholic University of Korea, Bucheon St.Mary's Hospital, Bucheon-si
  - Seoul National University Bundang Hospital, Seongnam
  - Kyung Hee University Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Soonchunhyang University Hospital Seoul, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (22):
  - Hospital General Universitario de Alicante, Alicante
  - Hospital del Mar, Barcelona
  - Hospital Universitari Vall D Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital de Basurto, Bilbao
  - Hospital Universitario Virgen de la Arrixaca, El Palmar
  - Hospital de Galdakao, Galdakao
  - Hospital Universitari de Girona Doctor Josep Trueta, Girona
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat
  - Hospital La Princesa, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Virgen de la Victoria, Málaga
  - Hospital Central de Asturias, Oviedo
  - Hospital Quirónsalud Madrid, Pozuelo de Alarcón
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Clínico de Santiago, Santiago de Compostela
  - Hospital Virgen del Rocío, Seville
  - Hospital Nuestra Señora de Valme, Seville
- Akademiska sjukhuset, Uppsala, Sweden
- Switzerland (2):
  - Universitätsspital Basel, Basel
  - University Hospital Bern, Bern
- Taiwan (5):
  - Chang-Hua Christian Hospital, Changhua
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - NCKUH, Tainan
  - Taipei Veterans General Hospital, Taipei
- Thailand (6):
  - Siriraj Hospital, Bangkok Noi
  - Songklanagarind Hospital, Hat Yai
  - Srinagarind Hospital, Khon Kaen
  - Central Chest Institute of Thailand, Muang
  - Maharat Nakhonchiangmai Hospital, Muang
  - Ramathibodi Hospital, Ratchatewi
- Turkey (Türkiye) (6):
  - Gulhane Training and Research Hospital, Ankara
  - Ankara Universitesi Tip Fakultesi, Ankara
  - Akdeniz Universitesi Tip Fakultesi -ANTALYA-33606, Antalya
  - Uludag Universitesi Tip Fakultesi, Bursa
  - Istanbul Universitesi Istanbul Tip Fakultesi, Istanbul
  - Gazi Universitesi Tip Fakultesi, Yenimahalle/ANKARA
- United Kingdom (13):
  - Aberdeen Royal Infirmary, Aberdeen
  - Queen Elizabeth Hospital Birmingham, Birmingham
  - Southmead Hospital, Bristol
  - Royal Infirmary of Edinburgh, Edinburgh
  - Royal Devon and Exeter Hospital, Wonford, Exeter
  - Royal Lancaster Infirmary, Lancaster
  - St James's University Hospital, Leeds
  - Guy's Hospital, London
  - Royal Brompton Hospital, London
  - Altnagelvin Area Hospital, Londonderry
  - Wythenshawe Hospital, Manchester
  - Churchill Hospital, Oxford
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Wuyts WA, Richeldi L, Assassi S, Azuma A, Cottin V, Hoffmann-Vold AM, Kreuter M, Oldham JM, Martinez FJ, Valenzuela C, Wijsenbeek MS, Kanakapura M, James A, Weimann G, Drzewuski C, Coeck C, Maher TM. Design of an open-label extension trial of nerandomilast (BI 1015550) in patients with idiopathic pulmonary fibrosis and progressive pulmonary fibrosis (FIBRONEER-ON). BMC Pulm Med. 2025 Dec 4;26(1):10. doi: 10.1186/s12890-025-03973-7. PMID 41345848
- [Derived] Maher TM, Assassi S, Azuma A, Cottin V, Hoffmann-Vold AM, Kreuter M, Oldham JM, Richeldi L, Valenzuela C, Wijsenbeek MS, Clerisme-Beaty E, Coeck C, Gu H, Ritter I, Schlosser A, Stowasser S, Voss F, Weimann G, Zoz DF, Martinez FJ; FIBRONEER-ILD Trial Investigators. Nerandomilast in Patients with Progressive Pulmonary Fibrosis. N Engl J Med. 2025 Jun 12;392(22):2203-2214. doi: 10.1056/NEJMoa2503643. Epub 2025 May 19. PMID 40388329
- [Derived] Maher TM, Assassi S, Azuma A, Cottin V, Hoffmann-Vold AM, Kreuter M, Oldham JM, Richeldi L, Valenzuela C, Wijsenbeek MS, Coeck C, Schlecker C, Voss F, Wachtlin D, Martinez FJ. Design of a phase III, double-blind, randomised, placebo-controlled trial of BI 1015550 in patients with progressive pulmonary fibrosis (FIBRONEER-ILD). BMJ Open Respir Res. 2023 Sep;10(1):e001580. doi: 10.1136/bmjresp-2022-001580. PMID 37709661
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multi-centre, multi-national, prospective, randomised, placebo-controlled, double-blind clinical trial, including a treatment period of at least 52 weeks, and a 1-week follow-up period in patients with progressive pulmonary fibrosis.
  The trial comprised two parts: Treatment Period A lasted up to 52 weeks post-randomisation, followed by Treatment Period B in which patients continued randomised blinded treatment for a variable duration.
Pre-assignment Details: All participants were screened for eligibility prior to participation in the trial. Participants attended a specialist site which ensured that they (the participants) strictly met all inclusion and none of the exclusion criteria. Participants were not to be allocated to a treatment sequence if any of the entry criteria were violated.
Period: Overall Study
Arm/Group | Placebo | Nerandomilast 9 mg | Nerandomilast 18 mg
Started (Randomized to treatment) | 393 | 393 | 392
Treated | 392 | 393 | 391
Completed treatment up to 52 weeks | 317 | 318 | 311
Completed (Completed treatment over the whole trial) | 271 | 283 | 272
Not Completed | 122 | 110 | 120
Not completed — Other than listed | 40 | 26 | 27
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Withdrawal by Subject | 30 | 34 | 42
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Adverse Event | 49 | 49 | 48
Not completed — Lack of Efficacy | 2 | 0 | 1
Not completed — Not treated | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): This patient set included all randomised patients who received at least one dose of study drug. The FAS was used for baseline demographics and characteristics, protocol deviations, and all efficacy analyses, in which patients were analysed as their randomised treatment group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Nerandomilast 9 mg | Nerandomilast 18 mg | Total
Number analyzed (Participants) | 392 | 393 | 391 | 1176
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.6 (10.3) | 66.5 (9.8) | 66.0 (9.8) | 66.4 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 161 | 190 | 171 | 522
  Male | 231 | 203 | 220 | 654
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 53 | 60 | 57 | 170
  Not Hispanic or Latino | 339 | 333 | 334 | 1006
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 6 | 2 | 13
  Asian | 149 | 155 | 143 | 447
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 7 | 3 | 6 | 16
  White | 226 | 224 | 235 | 685
  More than one race | 5 | 5 | 5 | 15
  Unknown or Not Reported | 0 | 0 | 0 | 0
Forced vital capacity (FVC) at baseline [Mean (Standard Deviation); unit: Milliliters (mL)] | 2353.6 (766.2) | 2325.5 (767.6) | 2381.4 (722.8) | 2353.4 (752.3)

OUTCOME MEASURES:

1. Secondary Outcome: Key Secondary Endpoint: Time to First Occurrence of Any of the Components of the Composite Endpoint: Time to First Acute ILD Exacerbation, First Hospitalisation for Respiratory Cause, or Death (Whichever Occurred First) Over the Duration of the Trial
Description: Time to first occurrence of any of the components of the composite endpoint - acute interstitial lung disease (ILD) exacerbation, first hospitalisation for respiratory cause, or death (whichever occurred first) - is reported as the number of participants who experienced any of these events during the trial.
  Acute exacerbation of ILD describes an acute, clinically significant, respiratory deterioration characterized by evidence of new widespread alveolar abnormality with all of the following: Acute worsening or development of dyspnea typically with less than 1 month duration, computed tomography with new bilateral ground-glass opacity and/or consolidation superimposed on a background pattern consistent with fibrosing ILD, and deterioration not fully explained by cardiac failure or fluid overload.
  If more than one component occurred on the same day, the patient was counted under the first event according to the following hierarchy: acute ILD exacerbation, hospitalization, death.
Time Frame: From first administration of trial drug (Nerandomilast or Placebo) till end of study, up to 26.2 months.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Nerandomilast 9 mg | Nerandomilast 18 mg
Number analyzed (Participants) | 392 | 393 | 391
Participants
  Acute ILD exacerbation as first event | 44 | 34 | 30
  Hospitalisation for respiratory cause as first event | 82 | 70 | 74
  Death as first event | 17 | 12 | 9
Statistical Analysis 1: Comparison: Placebo vs Nerandomilast 9 mg; The hazard ratio (HR) was estimated using a Cox proportional hazards model with treatment, baseline intake of AF (nintedanib) treatment, baseline HRCT pattern, age (continuous), baseline FVC % predicted, and baseline DLCO % predicted (corrected for hemoglobin) as covariates. Breslow's method was applied for tied event times. A two-sided p-value from the Wald test assessed the treatment effect. P-values were not adjusted for multiplicity; Test type: Superiority; p = 0.0507, Regression, Cox; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.61 to 1.00]
Statistical Analysis 2: Comparison: Placebo vs Nerandomilast 18 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0395, Regression, Cox; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.60 to 0.99]

2. Secondary Outcome: Time to First Acute ILD Exacerbation or Death Over the Duration of the Trial
Description: Time to first acute ILD exacerbation or death over the duration of the trial is reported as the number of patients who experienced either event. Acute exacerbation of ILD describes an acute, clinically significant, respiratory deterioration characterized by evidence of new widespread alveolar abnormality with all of the following: Acute worsening or development of dyspnea typically with less than 1 month duration, computed tomography with new bilateral ground-glass opacity and/or consolidation superimposed on a background pattern consistent with fibrosing ILD, and deterioration not fully explained by cardiac failure or fluid overload.
  If more than one component occurred on the same day, the patient was counted under the first event according to the following hierarchy: acute IPF exacerbation followed by death.
Time Frame: From first administration of trial drug (Nerandomilast or Placebo) till end of study, up to 26.2 months.
Population: Full Analysis Set (FAS): This patient set included all randomized patients who received at least one dose of study drug. The FAS was used for baseline demographics and characteristics, protocol deviations, and all efficacy analyses, in which patients were analyzed as their randomized treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Nerandomilast 9 mg | Nerandomilast 18 mg
Number analyzed (Participants) | 392 | 393 | 391
Participants
  Acute ILD exacerbation | 57 | 46 | 35
  Death | 40 | 24 | 24
Statistical Analysis 1: Comparison: Placebo vs Nerandomilast 9 mg; Analysis performed using a Cox proportional hazards model that included baseline antifibrotic therapy (AF group vs non-AF group), baseline HRCT pattern, age, baseline FVC % predicted, baseline diffusing capacity of the lungs for carbon monoxide (DLCO) % predicted (corrected for Hb) and treatment as covariates; Test type: Superiority; p = 0.0258, Regression, Cox; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.51 to 0.96]
Statistical Analysis 2: Comparison: Placebo vs Nerandomilast 18 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0017, Regression, Cox; Hazard Ratio (HR) = 0.59, 95% CI 2-sided [0.43 to 0.82]

3. Secondary Outcome: Time to Hospitalisation for Respiratory Cause or Death Over the Duration of the Trial
Description: Time to hospitalisation for respiratory cause or death over the duration of the trial is reported as the number of participants who experienced either event. Hospitalizations due to respiratory causes were recorded on a specific non-elective hospitalization CRF page. This page captured the hospitalization date, confirmation of a respiratory cause, and the primary admission diagnosis. Time to death was based either on the date of death on the adverse event (AE) report for patients with AEs leading to death or was based on the information from the vital status assessment.
Time Frame: From first administration of trial drug (Nerandomilast or Placebo) till end of study, up to 26.2 months.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Nerandomilast 9 mg | Nerandomilast 18 mg
Number analyzed (Participants) | 392 | 393 | 391
Participants
  Hospitalization for respiratory cause | 113 | 90 | 94
  Death | 18 | 13 | 9
Statistical Analysis 1: Comparison: Placebo vs Nerandomilast 9 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0237, Regression, Cox; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.57 to 0.96]
Statistical Analysis 2: Comparison: Placebo vs Nerandomilast 18 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0427, Regression, Cox; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.59 to 0.99]

4. Primary Outcome: Absolute Change From Baseline in Forced Vital Capacity (FVC) in Milliliters [mL] at Week 52
Description: The absolute change from baseline in forced vital capacity (FVC) in milliliters [mL] at Week 52 is reported. The absolute change from baseline in FVC was analyzed by a restricted maximum likelihood (REML)-based mixed model with repeated measurements (MMRM) comparing the change from baseline in FVC at Week 52 between treatment groups. The analysis included the fixed, categorical effects of treatment, baseline intake of antifibrotic (AF) treatment, and baseline High-resolution Computed Tomography (HRCT) pattern at each visit, as well as the fixed continuous effects of baseline FVC value at each visit. Visits were treated as a repeated measure with an unstructured covariance structure used to model within-patient measurements.
Time Frame: The MMRM model is a longitudinal analysis, and it incorporated FVC measurements change from baseline at Week 1, Week 2, Week 6, Week 12, Week 18, Week 26, Week 36, Week 44 and Week 52. Data presented is the FVC adjusted change from baseline at Week 52.
Population: Full Analysis Set (FAS): This patient set included all randomized patients who received at least one dose of study drug. The FAS was used for baseline demographics and characteristics, protocol deviations, and all efficacy analyses, in which patients were analyzed as their randomized treatment group. Only patients with baseline measurement and at least one post-baseline measurement were included.
Measure: Least Squares Mean (95% Confidence Interval); unit: Milliliters (mL)
Arm/Group | Placebo | Nerandomilast 9 mg | Nerandomilast 18 mg
Number analyzed (Participants) | 391 | 390 | 390
Milliliters (mL) | -165.77 [-190.52 to -141.03] | -84.64 [-109.63 to -59.65] | -98.59 [-123.74 to -73.44]
Statistical Analysis 1: Comparison: Placebo vs Nerandomilast 9 mg; Based on a Mixed Model for Repeated Measures (MMRM), with fixed, categorical effects of treatment at each visit, baseline antifibrotic therapy at each visit, baseline HRCT pattern at each visit, the fixed continuous effects of baseline FVC [mL] at each visit and unstructured covariance for repeated measures. Baseline antifibrotic therapy and HRCT pattern as entered in the CRF pages were used as covariates; Test type: Superiority; p < 0.0001, Mixed Models Analysis; The Kenward-Roger method estimated denominator degrees of freedom and adjusted standard errors; tests used two-sided α per multiple testing strategy; Mean Difference (Net) = 81.14, 95% CI 2-sided [45.95 to 116.32] — Adjusted mean difference in FVC change from baseline at Week 52 between the Nerandomilast 9 mg group and the Placebo group
Statistical Analysis 2: Comparison: Placebo vs Nerandomilast 18 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0002, Mixed Models Analysis; [statistical method as in outcome 4, analysis 1]; Mean Difference (Net) = 67.18, 95% CI 2-sided [31.91 to 102.46] — Adjusted mean difference in FVC change from baseline at Week 52 between the Nerandomilast 18 mg group and the Placebo group

5. Secondary Outcome: Time to Death Over the Duration of the Trial
Description: Time to death over the duration of the trial is reported as the number of participants who died.
  Time to death was based either on the date of death on the AE report for patients with AEs leading to death or based on the information from the vital status assessment.
Time Frame: From first administration of trial drug (Nerandomilast or Placebo) till end of study, up to 26.2 months.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Nerandomilast 9 mg | Nerandomilast 18 mg
Number analyzed (Participants) | 392 | 393 | 391
Participants | 64 | 36 | 34
Statistical Analysis 1: Comparison: Placebo vs Nerandomilast 9 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0017, Regression, Cox; Hazard Ratio (HR) = 0.51, 95% CI 2-sided [0.34 to 0.78]
Statistical Analysis 2: Comparison: Placebo vs Nerandomilast 18 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0018, Regression, Cox; Hazard Ratio (HR) = 0.51, 95% CI 2-sided [0.34 to 0.78]

6. Secondary Outcome: Absolute Change From Baseline in Forced Vital Capacity (FVC) Percent (%) Predicted at Week 52
Description: Absolute change from baseline in forced vital capacity (FVC) percent (%) predicted at Week 52 is reported.
  Analysis was based on a Mixed Model for Repeated Measures (MMRM), with fixed, categorical effects of treatment at each visit, baseline antifibrotic therapy at each visit, baseline HRCT pattern at each visit, the fixed continuous effects of baseline FVC [% pred] at each visit and unstructured covariance for repeated measures. Baseline antifibrotic therapy and HRCT pattern as entered in the CRF pages were used as covariates.
Time Frame: The MMRM model is a longitudinal analysis, and it incorporated FVC % predicted change from baseline at Week 1, Week 2, Week 6, Week 12, Week 18, Week 26, Week 36, Week 44 and Week 52. Data presented is change from baseline in FVC % predicted at Week 52.
Population: Full Analysis Set (FAS): This patient set included all randomized patients who received at least one dose of study drug. The FAS was used for baseline demographics and characteristics, protocol deviations, and all efficacy analyses, in which patients were analyzed as their randomized treatment group.
  Only participants with baseline measurement and at least one post-baseline measurement were included.
Measure: Least Squares Mean (95% Confidence Interval); unit: FVC percent predicted
Arm/Group | Placebo | Nerandomilast 9 mg | Nerandomilast 18 mg
Number analyzed (Participants) | 360 | 348 | 344
FVC percent predicted | -4.88 [-5.61 to -4.15] | -2.69 [-3.43 to -1.95] | -2.94 [-3.68 to -2.19]
Statistical Analysis 1: Comparison: Placebo vs Nerandomilast 9 mg; Based on MMRM, with fixed, categorical effects of treatment at each visit, baseline antifibrotic therapy at each visit, baseline HRCT pattern at each visit, the fixed continuous effects of baseline FVC [% pred] at each visit and unstructured covariance for repeated measures. Baseline antifibrotic therapy and HRCT pattern as entered in the CRF pages were used as covariates; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Net) = 2.19, 95% CI 2-sided [1.15 to 3.23] — The adjusted mean difference represents the model-estimated difference in predicted Forced Vital Capacity % between the Nerandomilast 9 mg group and the Placebo group at Week 52
Statistical Analysis 2: Comparison: Placebo vs Nerandomilast 18 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.0003, Mixed Models Analysis; Mean Difference (Net) = 1.94, 95% CI 2-sided [0.90 to 2.98] — The adjusted mean difference represents the model-estimated difference in predicted Forced Vital Capacity % between the Nerandomilast 18 mg group and the Placebo group at Week 52

7. Secondary Outcome: Time to Absolute Decline in Forced Vital Capacity (FVC) % Predicted of >10% From Baseline or Death Over the Duration of the Trial
Description: The time to absolute decline of more than 10% from baseline in forced vital capacity (FVC) percent predicted, or death, over the duration of the trial is reported as the number of participants who experienced either event.
  If multiple components occurred on the day of first event, then the patient was only counted in the first component based on the following hierarchy: absolute decline in FVC % predicted of > 10% followed by death.
Time Frame: From first administration of trial drug (Nerandomilast or Placebo) till end of study, up to 26.2 months.
Population: Full Analysis Set (FAS): This patient set includes all randomised patients who received at least one dose of study drug. The FAS was used for baseline demographics and characteristics, protocol deviations, and all efficacy analyses, in which patients were analysed as their randomised treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Nerandomilast 9 mg | Nerandomilast 18 mg
Number analyzed (Participants) | 392 | 393 | 391
Participants
  Absolute decline in FVC % predicted of > 10% | 130 | 95 | 100
  Death | 39 | 30 | 24
Statistical Analysis 1: Comparison: Placebo vs Nerandomilast 9 mg; Analysis was performed using a Cox proportional hazards regression model that included baseline use of antifibrotic therapy (antifibrotic group vs non-antifibrotic group), baseline HRCT pattern, age, baseline forced vital capacity (FVC) percentage predicted, baseline diffusing capacity of the lungs for carbon monoxide (DLCO) percentage predicted (corrected for hemoglobin levels), and treatment group as covariates; Test type: Superiority; p = 0.0018, Regression, Cox; Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.54 to 0.87]
Statistical Analysis 2: Comparison: Placebo vs Nerandomilast 18 mg; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.0038, Regression, Cox; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.56 to 0.89]

8. Secondary Outcome: Absolute Change From Baseline in Diffusing Capacity of the Lungs for Carbon Monoxide (DLCO) % Predicted (Corrected for Hb) at Week 52
Description: The absolute change from baseline in Diffusing Capacity of the Lungs for Carbon Monoxide percent predicted (corrected for hemoglobin, Hb) at Week 52 is reported.. Analysis was based on a Mixed Model for Repeated Measures (MMRM), with fixed, categorical effects of treatment at each visit, baseline antifibrotic therapy at each visit, baseline HRCT pattern at each visit, the fixed continuous effects of baseline DLCO [% pred] at each visit and unstructured covariance for repeated measures. Baseline antifibrotic therapy and HRCT pattern as entered in the CRF pages were used as covariates.
Time Frame: The MMRM model is a longitudinal analysis and it incorporated DLCO measurements from baseline (Week -8 to Week -1) and Week 12, Week 26, and Week 52. The data represent the adjusted Least Square Means for change from baseline at Week 52.
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: DLCO percent (%) predicted
Arm/Group | Placebo | Nerandomilast 9 mg | Nerandomilast 18 mg
Number analyzed (Participants) | 321 | 316 | 311
DLCO percent (%) predicted | -2.48 [-3.89 to -1.07] | -3.38 [-4.80 to -1.96] | -2.97 [-4.40 to -1.53]
Statistical Analysis 1: Comparison: Placebo vs Nerandomilast 9 mg; Analysis was based on a Mixed Model for Repeated Measures (MMRM), which included fixed, categorical effects of treatment, baseline use of antifibrotic therapy, and the fixed continuous effects of baseline DLCO [% pred] at each visit. An unstructured covariance structure was used to model repeated measures within patients. Baseline use of antifibrotic therapy, as recorded in the concomitant medication case report form page (CRF), was included as a covariate; Test type: Superiority; p = 0.3793, Mixed Models Analysis; Mean Difference (Net) = -0.90, 95% CI 2-sided [-2.90 to 1.11] — The adjusted mean difference represents the model-estimated difference in DLCO [% pred] between the Nerandomilast 9 mg group and the Placebo group at Week 52
Statistical Analysis 2: Comparison: Placebo vs Nerandomilast 18 mg; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.6354, Mixed Models Analysis; Mean Difference (Net) = -0.49, 95% CI 2-sided [-2.50 to 1.53] — The adjusted mean difference represents the model-estimated difference in DLCO [% pred] between the Nerandomilast 18 mg group and the Placebo group at Week 52

9. Secondary Outcome: Time to Absolute Decline in Diffusing Capacity of the Lungs for Carbon Monoxide (DLCO) Percentage Predicted by More Than 15% From Baseline or Death, Measured Over the Duration of the Trial
Description: Time to absolute decline in Diffusing Capacity of the Lungs for Carbon Monoxide (DLCO) percentage predicted by more than 15% from baseline or death, measured over the duration of the trial is reported as the number of participants who experienced either event. The Predicted DLCO value was corrected for hemoglobin (Hb). If more than one component occurred on the same day, the patient was counted under the first event according to the hierarchy: Absolute decline in DLCO % predicted of > 15%, followed by Death.
Time Frame: From first administration of trial drug (Nerandomilast or Placebo) till end of study, up to 26.2 months.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Nerandomilast 9 mg | Nerandomilast 18 mg
Number analyzed (Participants) | 392 | 393 | 391
Participants
  Absolute decline in DLCO % predicted of > 15% | 49 | 53 | 52
  Death | 58 | 35 | 32
Statistical Analysis 1: Comparison: Placebo vs Nerandomilast 9 mg; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.2967, Regression, Cox; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.65 to 1.14]
Statistical Analysis 2: Comparison: Placebo vs Nerandomilast 18 mg; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.4815, Regression, Cox; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.68 to 1.20]

10. Secondary Outcome: Absolute Change From Baseline in Living With Pulmonary Fibrosis (L-PF) Symptoms Dyspnea Domain Score at Week 52
Description: The absolute change from baseline in Living with Pulmonary Fibrosis (L-PF) Symptoms Dyspnea domain score at Week 52 is reported. The Living with Pulmonary Fibrosis (L-PF) questionnaire is a 44-item tool consisting of two modules: Symptoms (23 items) and Impacts (21 items). The Symptoms module yields three domain scores: Dyspnoea, Cough, and Fatigue, as well as a Total Symptoms score. Scoring is based on the mean of item ratings within each domain, multiplied by 100. Scores range from 0 to 100, with higher scores indicating greater impairment.
  This endpoint was analyzed using a Mixed Model for Repeated Measures (MMRM). The model included fixed effects for treatment, baseline antifibrotic therapy, baseline HRCT pattern, and fixed continuous effect of baseline L-PF dyspnea score at each visit, with an unstructured covariance for repeated measures. Baseline antifibrotic therapy and HRCT pattern as entered in the CRF pages were covariates.
Time Frame: The MMRM model is a longitudinal analysis and it incorporated L-PF measurements from baseline (Week -8 to Week -1) and Week 12, Week 26, Week 36, Week 44 and Week 52. The data represent the adjusted Least Square Means for change from baseline at Week 52.
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Placebo | Nerandomilast 9 mg | Nerandomilast 18 mg
Number analyzed (Participants) | 331 | 329 | 328
Score on a scale | 5.75 [4.04 to 7.46] | 4.87 [3.15 to 6.58] | 4.48 [2.76 to 6.20]
Statistical Analysis 1: Comparison: Placebo vs Nerandomilast 9 mg; Analysis was based on a Based on Mixed Model for Repeated Measures (MMRM), with fixed, categorical effects of treatment at each visit, baseline antifibrotic therapy at each visit, baseline HRCT pattern at each visit, the fixed continuous effects of baseline L-PF Dyspnea score at each visit and unstructured covariance for repeated measures. Baseline antifibrotic therapy and HRCT pattern as entered in the CRF pages were used as covariates; Test type: Superiority; p = 0.4748, Mixed Models Analysis; Mean Difference (Net) = -0.88, 95% CI 2-sided [-3.30 to 1.54] — The adjusted mean difference represents the model-estimated difference in symptom change (L-PF Dyspnea score) between the Nerandomilast 9mg group and the Placebo group at Week 52
Statistical Analysis 2: Comparison: Placebo vs Nerandomilast 18 mg; Analysis was based on a Mixed Model for Repeated Measures (MMRM), with fixed, categorical effects of treatment at each visit, baseline antifibrotic therapy at each visit, baseline HRCT pattern at each visit, the fixed continuous effects of baseline L-PF Dyspnea score at each visit and unstructured covariance for repeated measures. Baseline antifibrotic therapy and HRCT pattern as entered in the CRF pages were used as covariates; Test type: Superiority; p = 0.3042, Mixed Models Analysis; Mean Difference (Net) = -1.27, 95% CI 2-sided [-3.69 to 1.15] — The adjusted mean difference represents the model-estimated difference in symptom change (L-PF Dyspnea score) between the Nerandomilast 18 mg group and the Placebo group at Week 52

11. Secondary Outcome: Absolute Change From Baseline in Living With Pulmonary Fibrosis (L-PF) Symptoms Cough Domain Score at Week 52
Description: The absolute change from baseline in the L-PF Cough domain score at Week 52 is reported. The Living with Pulmonary Fibrosis (L-PF) questionnaire is a 44-item tool consisting of two modules: Symptoms (23 items) and Impacts (21 items). The Symptoms module yields three domain scores: Dyspnea, Cough, and Fatigue, as well as a Total Symptoms score. Scoring is based on the mean of item ratings within each domain, multiplied by 100. Scores range from 0 to 100, with higher scores indicating greater impairment.
  This endpoint was analyzed using a Mixed Model for Repeated Measures (MMRM). The model included fixed effects for treatment, baseline antifibrotic therapy, baseline HRCT pattern, and fixed continuous effect of baseline L-PF dyspnea score at each visit, with an unstructured covariance for repeated measures. Baseline antifibrotic therapy and HRCT pattern as entered in the CRF pages were covariates.
Time Frame: as for outcome 10
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Placebo | Nerandomilast 9 mg | Nerandomilast 18 mg
Number analyzed (Participants) | 331 | 328 | 328
Score on a scale | 3.05 [0.79 to 5.31] | 1.17 [-1.09 to 3.44] | 3.19 [0.92 to 5.46]
Statistical Analysis 1: Comparison: Placebo vs Nerandomilast 9 mg; Analysis was based on a Mixed Model for Repeated Measures (MMRM), with fixed, categorical effects of treatment at each visit, baseline antifibrotic therapy at each visit, baseline HRCT pattern at each visit, the fixed continuous effects of baseline L-PF Cough score at each visit and unstructured covariance for repeated measures. Baseline antifibrotic therapy and HRCT pattern as entered in the CRF pages were used as covariates; Test type: Superiority; p = 0.2506, Mixed Models Analysis; Mean Difference (Net) = -1.88, 95% CI 2-sided [-5.08 to 1.33], Standard Error of Mean 1.63 — The adjusted mean difference represents the model-estimated difference in symptom change (L-PF Cough score) between the Nerandomilast 9 mg group and the Placebo group at Week 52
Statistical Analysis 2: Comparison: Placebo vs Nerandomilast 18 mg; [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p = 0.9311, Mixed Models Analysis; Mean Difference (Net) = 0.14, 95% CI 2-sided [-3.07 to 3.35] — The adjusted mean difference represents the model-estimated difference in symptom change (L-PF Cough score) between the Nerandomilast 18 mg group and the Placebo group at Week 52

12. Secondary Outcome: Absolute Change From Baseline in Living With Pulmonary Fibrosis (L-PF) Symptoms Fatigue Domain Score at Week 52
Description: The absolute change from baseline in the L-PF Fatigue domain score at Week 52 is reported. The Living with Pulmonary Fibrosis (L-PF) questionnaire is a 44-item tool consisting of two modules: Symptoms (23 items) and Impacts (21 items). The Symptoms module yields three domain scores: Dyspnea, Cough, and Fatigue, as well as a Total Symptoms score. Scoring is based on the mean of item ratings within each domain, multiplied by 100. Scores range from 0 to 100, with higher scores indicating greater impairment.
  This endpoint was analyzed using a Mixed Model for Repeated Measures (MMRM). The model included fixed effects for treatment, baseline antifibrotic therapy, and baseline HRCT pattern at each visit, and fixed continuous effect of baseline L-PF Fatigue score at each visit, with an unstructured covariance for repeated measures. Baseline antifibrotic therapy and HRCT pattern as entered in the CRF pages were covariates.
Time Frame: as for outcome 10
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Placebo | Nerandomilast 9 mg | Nerandomilast 18 mg
Number analyzed (Participants) | 331 | 329 | 327
Score on a scale | 2.95 [1.18 to 4.73] | 3.01 [1.23 to 4.78] | 3.89 [2.11 to 5.68]
Statistical Analysis 1: Comparison: Placebo vs Nerandomilast 9 mg; Analysis was based on a Mixed Model for Repeated Measures (MMRM), with fixed, categorical effects of treatment at each visit, baseline antifibrotic therapy at each visit, baseline HRCT pattern at each visit, the fixed continuous effects of baseline L-PF Fatigue score at each visit and unstructured covariance for repeated measures. Baseline antifibrotic therapy and HRCT pattern as entered in the CRF pages were used as covariates; Test type: Superiority; p = 0.9668, Mixed Models Analysis; Mean Difference (Net) = 0.05, 95% CI 2-sided [-2.46 to 2.57] — The adjusted mean difference represents the model-estimated difference in symptom change (L-PF Fatigue score) between the Nerandomilast 9mg group and the Placebo group at Week 52
Statistical Analysis 2: Comparison: Placebo vs Nerandomilast 18 mg; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p = 0.4644, Mixed Models Analysis; Mean Difference (Net) = 0.94, 95% CI 2-sided [-1.58 to 3.46] — The adjusted mean difference represents the model-estimated difference in symptom change (L-PF Fatigue score) between the Nerandomilast 18 mg group and the Placebo group at Week 52

ADVERSE EVENTS:
Time Frame: Serious and Other adverse events, All-cause mortality: From first drug administration until end of trial, plus a residual effect period of 7 days, up to 26.4 months.
Description: Treated Set (TS): This patient set included all randomized patients who received at least one dose of study drug.
Arm/Group | Placebo | Nerandomilast 9 mg | Nerandomilast 18 mg
All-Cause Mortality (participants affected / at risk) | 64/392 | 36/393 | 34/391
Serious Adverse Events (participants affected / at risk) | 198/392 | 174/393 | 182/391
Other Adverse Events (participants affected / at risk) | 320/392 | 324/393 | 333/391
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=392) | Nerandomilast 9 mg (N=393) | Nerandomilast 18 mg (N=391)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 2
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Acute left ventricular failure (Cardiac disorders) | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 1 | 3
Angina pectoris (Cardiac disorders) | 0 | 1 | 3
Angina unstable (Cardiac disorders) | 0 | 1 | 3
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 3 | 5
Atrial flutter (Cardiac disorders) | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 3 | 2 | 0
Cardiac failure (Cardiac disorders) | 5 | 2 | 5
Cardiac failure acute (Cardiac disorders) | 3 | 0 | 0
Cardiac failure chronic (Cardiac disorders) | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 1 | 0
Conduction disorder (Cardiac disorders) | 0 | 1 | 0
Cor pulmonale acute (Cardiac disorders) | 1 | 1 | 0
Cor pulmonale chronic (Cardiac disorders) | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 2 | 6 | 1
Coronary artery occlusion (Cardiac disorders) | 0 | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 2 | 0
Heart failure with preserved ejection fraction (Cardiac disorders) | 0 | 1 | 0
Heart failure with reduced ejection fraction (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 2 | 3
Myocardial injury (Cardiac disorders) | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1
Prinzmetal angina (Cardiac disorders) | 0 | 0 | 1
Right ventricular failure (Cardiac disorders) | 1 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 1 | 0
Porokeratosis (Congenital, familial and genetic disorders) | 1 | 0 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 1 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 | 0 | 0
Cataract (Eye disorders) | 1 | 0 | 1
Cataract cortical (Eye disorders) | 0 | 0 | 1
Cataract subcapsular (Eye disorders) | 1 | 0 | 0
Central serous chorioretinopathy (Eye disorders) | 0 | 1 | 0
Conjunctivochalasis (Eye disorders) | 0 | 0 | 1
Dry age-related macular degeneration (Eye disorders) | 0 | 1 | 0
Macular hole (Eye disorders) | 0 | 0 | 1
Macular rupture (Eye disorders) | 0 | 0 | 1
Ocular retrobulbar haemorrhage (Eye disorders) | 0 | 0 | 1
Retinal detachment (Eye disorders) | 1 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1
Acute abdomen (Gastrointestinal disorders) | 1 | 0 | 0
Chronic gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 0
Diverticular perforation (Gastrointestinal disorders) | 0 | 1 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 1
Gastric antral vascular ectasia (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 1
Gastritis erosive (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1
Ileus paralytic (Gastrointestinal disorders) | 0 | 1 | 0
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 1 | 2
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 1
Large intestinal stenosis (Gastrointestinal disorders) | 1 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 2 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0
Obstructive pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatic failure (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 2 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 2 | 1 | 0
Peptic ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Pneumoperitoneum (Gastrointestinal disorders) | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Rectal polyp (Gastrointestinal disorders) | 0 | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 2
Chest pain (General disorders) | 1 | 3 | 0
Condition aggravated (General disorders) | 54 | 41 | 27
Death (General disorders) | 6 | 5 | 6
Disease progression (General disorders) | 3 | 1 | 2
Fatigue (General disorders) | 1 | 1 | 0
General physical health deterioration (General disorders) | 0 | 1 | 1
Oedema peripheral (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Sudden cardiac death (General disorders) | 1 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0
Cholangitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 3 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 2 | 0 | 3
Congestive hepatopathy (Hepatobiliary disorders) | 0 | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 2 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 3 | 2 | 0
Suspected drug-induced liver injury (Hepatobiliary disorders) | 0 | 1 | 1
Anaphylactoid reaction (Immune system disorders) | 0 | 0 | 1
Anti-neutrophil cytoplasmic antibody positive vasculitis (Immune system disorders) | 0 | 1 | 0
Cell-mediated immune deficiency (Immune system disorders) | 0 | 1 | 0
Sarcoidosis (Immune system disorders) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0
Aspergillus infection (Infections and infestations) | 1 | 0 | 0
Atypical mycobacterial infection (Infections and infestations) | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 2 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 1
Bronchiolitis (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 2 | 1
Bronchitis bacterial (Infections and infestations) | 0 | 0 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 1 | 2
COVID-19 (Infections and infestations) | 9 | 7 | 6
COVID-19 pneumonia (Infections and infestations) | 0 | 1 | 4
Cellulitis (Infections and infestations) | 0 | 1 | 1
Citrobacter infection (Infections and infestations) | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 2 | 1 | 0
Epididymitis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 3 | 0 | 0
Haemophilus infection (Infections and infestations) | 0 | 1 | 1
Hepatitis E (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1
Infected cyst (Infections and infestations) | 0 | 0 | 1
Infection (Infections and infestations) | 3 | 0 | 0
Infectious pleural effusion (Infections and infestations) | 1 | 0 | 0
Infective exacerbation of bronchiectasis (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 3 | 2 | 6
Lower respiratory tract infection (Infections and infestations) | 1 | 2 | 4
Lower respiratory tract infection bacterial (Infections and infestations) | 0 | 0 | 1
Medical device site infection (Infections and infestations) | 0 | 0 | 1
Meningitis aseptic (Infections and infestations) | 1 | 0 | 0
Meningitis viral (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0
Ophthalmic herpes zoster (Infections and infestations) | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 0 | 1
Peritonsillar abscess (Infections and infestations) | 1 | 0 | 0
Pneumocystis jirovecii infection (Infections and infestations) | 1 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 32 | 37 | 35
Pneumonia aspiration (Infections and infestations) | 2 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 6 | 4 | 3
Pneumonia fungal (Infections and infestations) | 1 | 0 | 1
Pneumonia influenzal (Infections and infestations) | 0 | 3 | 0
Pneumonia necrotising (Infections and infestations) | 0 | 1 | 0
Pneumonia pneumococcal (Infections and infestations) | 2 | 0 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 1 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 1 | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 4 | 2
SARS-CoV-2 sepsis (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 2 | 5
Septic shock (Infections and infestations) | 1 | 3 | 2
Serratia infection (Infections and infestations) | 0 | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 2 | 1
Urinary tract infection (Infections and infestations) | 1 | 1 | 1
Viral infection (Infections and infestations) | 2 | 0 | 0
Accident (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Asbestosis (Injury, poisoning and procedural complications) | 1 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Comminuted fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Craniofacial fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 2 | 1 | 0
Kidney rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0
Scapula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skull fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 3 | 1 | 3
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
C-reactive protein increased (Investigations) | 0 | 1 | 0
ECG signs of myocardial ischaemia (Investigations) | 0 | 0 | 1
Heart rate increased (Investigations) | 0 | 1 | 0
Human metapneumovirus test positive (Investigations) | 1 | 0 | 0
Imaging procedure abnormal (Investigations) | 0 | 0 | 1
Influenza A virus test positive (Investigations) | 0 | 0 | 1
Influenza B virus test positive (Investigations) | 0 | 0 | 1
Mycobacterium tuberculosis complex test positive (Investigations) | 1 | 0 | 1
Oxygen saturation decreased (Investigations) | 1 | 0 | 0
Pneumocystis test positive (Investigations) | 0 | 1 | 0
Respiratory rate increased (Investigations) | 0 | 0 | 1
Streptococcus test positive (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1 | 0
Steroid diabetes (Metabolism and nutrition disorders) | 1 | 0 | 0
Antisynthetase syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Dermatomyositis (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Idiopathic inflammatory myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Jaw cyst (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Polymyositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Scleroderma (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Systemic scleroderma (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0
Adenosquamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 4
Benign anorectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Localised melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 4
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 4
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Carotid artery dissection (Nervous system disorders) | 0 | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 3 | 1 | 1
Cerebrovascular insufficiency (Nervous system disorders) | 0 | 0 | 1
Cubital tunnel syndrome (Nervous system disorders) | 0 | 0 | 1
Dementia (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0
Hypercapnic coma (Nervous system disorders) | 0 | 1 | 0
Hypertensive encephalopathy (Nervous system disorders) | 0 | 1 | 0
Lacunar infarction (Nervous system disorders) | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 1
Migraine with aura (Nervous system disorders) | 0 | 0 | 1
Sciatica (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1
Spondylitic myelopathy (Nervous system disorders) | 0 | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 3
Transient ischaemic attack (Nervous system disorders) | 1 | 2 | 2
Vagus nerve paralysis (Nervous system disorders) | 0 | 1 | 0
Vertebral artery stenosis (Nervous system disorders) | 0 | 1 | 0
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 0 | 1
Device loosening (Product issues) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 2 | 1 | 2
Delirium (Psychiatric disorders) | 1 | 1 | 4
Depression (Psychiatric disorders) | 2 | 2 | 1
Disorientation (Psychiatric disorders) | 1 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 2 | 1 | 3
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 4 | 1
Anuria (Renal and urinary disorders) | 0 | 1 | 0
Glomerulonephritis (Renal and urinary disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 1
Renal colic (Renal and urinary disorders) | 0 | 0 | 1
Renal cyst (Renal and urinary disorders) | 1 | 0 | 0
Adnexa uteri mass (Reproductive system and breast disorders) | 0 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 2 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 4
Alveolar proteinosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Choking (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 6 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypersensitivity pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 10 | 7 | 8
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 6
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 13 | 8 | 6
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 5
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 5 | 7 | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 15 | 9 | 12
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 14 | 10 | 10
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Vocal cord leukoplakia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Aortic dissection (Vascular disorders) | 0 | 1 | 0
Aortic thrombosis (Vascular disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 3 | 2 | 2
Hypertension (Vascular disorders) | 1 | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 2 | 0
Subclavian artery thrombosis (Vascular disorders) | 1 | 0 | 0
Varicose vein (Vascular disorders) | 0 | 1 | 0
Vasculitis (Vascular disorders) | 0 | 2 | 0
Vena cava thrombosis (Vascular disorders) | 0 | 1 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=392) | Nerandomilast 9 mg (N=393) | Nerandomilast 18 mg (N=391)
Diarrhoea (Gastrointestinal disorders) | 107 | 129 | 151
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 16 | 22 | 13
Nausea (Gastrointestinal disorders) | 30 | 36 | 50
Vomiting (Gastrointestinal disorders) | 28 | 22 | 27
Condition aggravated (General disorders) | 34 | 28 | 26
Fatigue (General disorders) | 27 | 24 | 25
Pyrexia (General disorders) | 27 | 13 | 19
Bronchitis (Infections and infestations) | 32 | 37 | 30
COVID-19 (Infections and infestations) | 57 | 48 | 54
Influenza (Infections and infestations) | 27 | 18 | 25
Nasopharyngitis (Infections and infestations) | 53 | 54 | 51
Pneumonia (Infections and infestations) | 23 | 24 | 30
Respiratory tract infection (Infections and infestations) | 20 | 27 | 30
Upper respiratory tract infection (Infections and infestations) | 71 | 51 | 55
Urinary tract infection (Infections and infestations) | 27 | 31 | 23
Weight decreased (Investigations) | 36 | 44 | 58
Decreased appetite (Metabolism and nutrition disorders) | 31 | 28 | 39
Arthralgia (Musculoskeletal and connective tissue disorders) | 22 | 30 | 34
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 16 | 27
Dizziness (Nervous system disorders) | 14 | 19 | 21
Headache (Nervous system disorders) | 27 | 18 | 33
Anxiety (Psychiatric disorders) | 50 | 46 | 53
Depression (Psychiatric disorders) | 54 | 45 | 51
Cough (Respiratory, thoracic and mediastinal disorders) | 63 | 59 | 68
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 39 | 40 | 42
Hypertension (Vascular disorders) | 14 | 16 | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-09-21): https://cdn.clinicaltrials.gov/large-docs/82/NCT05321082/Prot_000.pdf
  • Statistical Analysis Plan (2024-12-30): https://cdn.clinicaltrials.gov/large-docs/82/NCT05321082/SAP_001.pdf